CLINICAL TRIAL: NCT00892632
Title: A Pilot Study of Confocal Endomicroscopy for Biliary Strictures - Phase I
Brief Title: Confocal Endomicroscopy for Biliary Strictures -Phase I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult (slow) Enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Wallace, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-008669
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Biliary Stricture
Keywords: Biliary Strictures; Cholangiocarcinoma; ERCP
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 1. To compare confocal image characteristics of benign vs. malignant biliary strictures
  Interventions: Procedure: ERCP and Confocal imaging

INTERVENTIONS:
Procedure: ERCP and Confocal imaging — A major new advancement in cancer imaging is the development of a probe-based confocal endomicroscopy (pCLE) system capable of cellular and sub-cellular imaging of the biliary tree.

SUMMARY:
The investigators hypothesize that the confocal endomicroscopy imaging of the biliary strictures during ERCP will differentiate between benign and malignant strictures in vivo and has increased sensitivity compared to biliary brushing/biopsy, and that direct cholangioscopic guidance of pCLE is more accurate than fluoroscopic guidance.

DETAILED DESCRIPTION:
Despite recent advances in biliary imaging and biliary tissue acquisition, the diagnosis and tissue-confirmation in suspected malignant biliary obstruction remains challenging. Patients often undergo repeat endoscopic and cross sectional imaging procedures, and even surgical exploration to establish a diagnosis. A major new advancement in cancer imaging is the development of a probe-based confocal endomicroscopy (pCLE) system capable of cellular and sub-cellular imaging of the biliary tree. Preliminary data suggests that pCLE can accurately detect or exclude malignancy within otherwise indeterminate strictures. In this study, we propose to validate these preliminary findings and compare two methods of pCLE image acquisition that are important for clinical translation of the technology.

This is a Phase 1 Study: During this study, in vivo microscopic images of 10 benign (post-operative from know benign disease such as orthotopic liver transplant) and 10 malignant (cytology-positive) strictures will be obtained at ERCP. Patients clinical course will be followed and a composite gold standard will be used for comparison to pCLE. These confocal images of biliary lesions will be reviewed side by side, unblinded to the reference standard by the endoscopists. The basic image characteristics allowing distinction between benign and malignant tissue will be established (details of features noted and examined are below). We will also assess whether good quality images can be feasibly obtained without the cholangioscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Pre-ERCP: Age above 18; imaging consistent with stenosis/mass of the hilum/extra-hepatic bile duct with abnormal liver chemistry, or painless jaundice referred for ERCP.
* Evidence of biliary obstruction as defined by elevated direct bilirubin (> 1.5ULN) and dilation of the common or hepatic ducts > 8mm) on imaging studies.

Exclusion Criteria:

* Unwilling/unable to consent.
* Definite pancreatic mass on CT/MR.
* Allergy to Fluorescein.
* Pregnancy (patient who could be pregnant will undergo pregnancy testing as per routine care)
* Indwelling metal biliary stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Primary Aim: 1. To compare confocal image characteristics of benign vs. malignant biliary strictures. | one year

SECONDARY OUTCOMES:
Secondary Aim: 1. To compare the technical feasibility (percentage of images rated as adequate or better) and the quality of the images obtained via fluoroscopy-guided pCLE versus cholangioscopy-guided pCLE. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Wallace, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States